CLINICAL TRIAL: NCT05523804
Title: Patient Outcomes Following Interval and Delayed Cytoreductive Surgery in Advanced Ovarian Cancer: A GO SOAR Led Study (GO SOAR2)
Brief Title: Patient Outcomes Following Interval and Delayed Cytoreductive Surgery in Advanced Ovarian Cancer
Acronym: GO SOAR2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Grampian (Other Government)
Collaborators: University of Aberdeen (Other); Barts & The London NHS Trust (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Faiza Gaba, Principle Investigator, University of Aberdeen
Other Study IDs: 5719
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer
Keywords: survival; morbidity; cytoreduction; disparities
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- interval cytoreductive surgery: women with stage III-IV ovarian cancer, undergoing interval (after 3-4 cycles of chemotherapy) cytoreductive surgery
  Interventions: Procedure: interval cytoreductive surgery
- delayed cytoreductive surgery: women with stage III-IV ovarian cancer, undergoing delayed (>5 cycles of chemotherapy) cytoreductive surgery
  Interventions: Procedure: delayed cytoreductive surgery
- no surgery: women with stage III-IV ovarian cancer, undergoing >5 cycles of chemotherapy alone (no cytoreductive surgery)
  Interventions: Other: no surgery

INTERVENTIONS:
Procedure: interval cytoreductive surgery — cytoreductive surgery after 3-4 cycles of chemotherapy
  Groups: interval cytoreductive surgery
Procedure: delayed cytoreductive surgery — surgery after >5 cycles of chemotherapy
  Groups: delayed cytoreductive surgery
Other: no surgery — no cytoreductive surgery (>5 cycles of chemotherapy alone)
  Groups: no surgery

SUMMARY:
To compare patient outcomes following interval and delayed cytoreductive surgeries and no surgery (neoadjuvant chemotherapy alone) and international variations in access to cytoreductive surgeries in women with advanced stage ovarian cancer.

DETAILED DESCRIPTION:
Standard of care in patients with advanced ovarian cancer is primary cytoreductive surgery followed by chemotherapy. Neoadjuvant chemotherapy and interval cytoreductive surgery is an alternative in selected patients. Most data exist with interval cytoreductive surgery following 3-4 cycles of chemotherapy, however, some patients experience a delay. So far, the impact of delayed cytoreductive surgery (following >5 cycles of chemotherapy) on patient outcomes is poorly defined. There is also a paucity of data in women who undergo no surgery (>5 cycles of chemotherapy alone) and factors influencing international discrepancies in access to cytoreductive surgery.

ELIGIBILITY:
Inclusion Criteria:

Women with stage III-IV ovarian cancer, undergoing interval (after 3-4 cycles of chemotherapy) or delayed (>5 cycles of chemotherapy) cytoreductive surgeries or no cytoreductive surgery (>5 cycles of chemotherapy alone.

Exclusion Criteria:

Women undergoing recurrent cytoreductive surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: women with stage III-IV ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 15 years
  defined from date of diagnosis to date of death by any cause or loss to follow-up
progression free survival | 15 years
  defined from date of diagnosis to date of first recurrence
facilitator/barriers to access to cytoreductive surgery | 15 years
  topic guide interview questionnaire to be used to elicit factors aiding/preventing access to cytoreductive surgery internationally

SECONDARY OUTCOMES:
Post-operative morbidity | within 30 days from date of surgery
  as per Clavien-Dindo classification
Resectability rates | at time of surgery
  R0 = no visible disease, R1 = <10mm visible residual disease, R2 = >10mm visible residual disease

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Gaba F, Ash K, Blyuss O, Bizzarri N, Kamfwa P, Ramirez PT, Kotsopoulos IC, Chandrasekaran D, Gomes N, Butler J, Nobbenhuis M, Ind T, Heath O, Barton D, Jeyarajah A, Brockbank E, Lawrence A, Dilley J, Manchanda R, Phadnis S, Soar GO. Patient outcomes following interval and delayed cytoreductive surgery in advanced ovarian cancer: protocol for a multicenter, international, cohort study (Global Gynaecological Oncology Surgical Outcomes Collaborative). Int J Gynecol Cancer. 2022 Dec 5;32(12):1606-1610. doi: 10.1136/ijgc-2022-004101. PMID 36379595